CLINICAL TRIAL: NCT04874337
Title: In Nursing Students, The Effect of Disaster Nursing Training Program on General Disaster Preparedness Belief State, Disaster Response Self-Efficiency and Psychological Resilience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Kent University (Other)
Collaborators: Istanbul Aydın University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 58797649-050
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: General Disaster Preparedness Belief State; Disaster Response Self-Efficiency; Psychological Resilience; Nursing Students
Keywords: General Disaster Preparedness Belief State; Disaster Response Self-Efficiency; Psychological Resilience; Nursing Students
MeSH Terms: interventions — Disaster Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Disaster nursing and management training will be given to students using Jenning's Disaster Nursing and Management Model.
  Interventions: Other: Disaster nursing and management training will be given to students using Jenning's Disaster Nursing and Management Model.
- Control Group (No Intervention)

INTERVENTIONS:
Other: Disaster nursing and management training will be given to students using Jenning's Disaster Nursing and Management Model. — The subjects for the training program were prepared by the researchers by scanning the relevant literature. In particular, the ICN Framework of Disaster Nursing Competencies developed by the International Nurses Association (ICN) and the World Health Organization (WHO), the second is the universal standards that should be fundamental in nursing and midwifery education (Global Standards for the Initial Education of Professional Nurses and Midwives). The training program was conducted both theoretically and practically. The theoretical section is based on Jenning's disaster nursing management model. Investigator is a First and Emergency Aid instructor. In addition, support was received from an experienced psychologist and AFAD trainers who provided support to the victims of the Izmir earthquake during the training process. In this context, an 8-module training program was created.
  Arms: Experimental group

SUMMARY:
In order to respond correctly to disasters, medical teams must have the necessary training and sufficient equipment. However, in many countries, disaster nursing education is not adequately included in nursing curricula (Kalanlar and Kublai, 2015). This is seen as an important situation affecting the capacity of nurses to respond to disasters. In particular, it is emphasized that providing disaster nursing and management training to nurse students will have positive consequences for disaster-affected individuals and communities, such as reduced death rates, improved health services, and reduced disaster-related costs (Kalanlar and Kublai, 2015). For this reason, disaster preparation of both nurses and student nurses is important for combating disasters.

It has been reported that nursing students provide assistance in issues such as monitoring the physical and psychological health of disaster victims, improving hygiene, and health counseling, using the knowledge and skills acquired in vocational education (Kashiwaba and Okudera, 2014; Tomizawa et al., 2014). Some studies have shown that student nurses do not have sufficient knowledge and skills in disaster preparedness and response (Schmidt et al., 2011; Smithers et al., 2020). However, in most schools where the curricula of domestic nursing schools are examined, disaster nursing courses are conducted as electives rather than majors. Despite these limitations, nursing students tops the teams that have a key role in a potential disaster or disaster (Satoh et al., 2016). Therefore, groups that can contribute during disaster response must have sufficient knowledge and skills. Because the lack of experience during intervention leads to stress and fear of intervening in disasters, while the belief that it is adequately prepared for disaster situations increases confidence in intervening in disasters. To overcome the lack of experience in Disaster Response, Education that will provide insight into the reality of disaster response is important.

To achieve the goal of training medical personnel capable of disaster response, a variety of training methods are needed, such as not only in-depth theory training, but also Case-Based Learning and practice in simulated situations with a multidisciplinary approach. In this context, the education model that stands out in the literature is the disaster nursing and management model developed by Jening. Jenning's disaster nursing management model was developed directly for Nurse students and describes the nurse's duties at each stage of Disaster Management. It is a model developed to explain disaster nursing to students and to provide them with knowledge about disaster management. In this aspect, the model differs from other disaster management models (Jennings Sanders, 2004).

The aim of this research is to evaluate the impact of disaster nursing and management education given to students using Jenning's disaster nursing and management model on general disaster preparedness belief state, disaster response self-efficiency and psychological resilience of students.

ELIGIBILITY:
Inclusion Criteria:

Nursing students aged 18 and over, who volunteer for the study, do not have any communication problems, do not take first and emergency courses will be included in the study

Exclusion Criteria:

Withdraw from study, Declined to participate,

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
General Disaster Preparedness Belief Scale | 3 weeks
  The General Disaster Preparedness Belief Scale was developed in 2018 by Inal et al. The scale based on the Health Belief model measures belief in disaster preparedness. The scale, consisting of 31 items, has 6 sub-dimensions. These are self efficacy (8 items), cues to action (5 items), perceived susceptibility (6 items), perceived barriers (6 items), perceived benefits (3 items) and perceived severity (3 items). The scale has no breakpoint. Cronbach's alpha coefficient for the subscales ranged from 0.90 to 0.74. In the study, the cronbach alpha (α) value of the scale was found to be 0.81. The scale's scoring system is coded for each expression as (1) strongly disagree, (2) disagree, (3) disagree, (4) agree, (5) strongly agree. The minimum score is 31 points and the maximum is 155 points.
The Disaster Response Self-Efficacy Scale | 3 weeks
  The Disaster Response Self-Efficacy Scale was developed in 2017 by Hong-Yan Li et al. Validity and reliability studies of the Turkish form of the scale were conducted by Koca et al. (2018). It consisted of a total of 19 items and 3 sub-dimensions, and the answers were taken with a likert scale of 5.(1=no self-confidence, 2=basically no self-confidence, 3=some self-confidence, 4=basically self-confidence, 5 = full self-confidence). High scores indicate that disaster response self-sufficiency is high. The Cronbach alpha coefficient was 0.96. For on-site rescue competency, disaster psychological nursing competency, disaster role quality and adaptation competency subscales, it was 0.93.
Brief Resilience Scale (BRS) | 3 weeks
  This self-reporting instrument developed by Smith et al. (2008) to measure the psychological well-being of individuals. The Turkish adaptation and psychometric studies of the scale were performed by Tayfun Doğan on 295 university students (2015). Explanatory and confirmatory factor analyses showed that the scale had a single-factor structure. The high scores obtained from the scale after translating the items coded in reverse order in the scale (items 2, 4 and 6) indicate a high psychological strength. Factor analysis was performed to determine the construct validity of the scale. The factor loads related to the items were found to be between 0.68 and 0.91 (Doğan, 2015).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doğan T. Kısa Psikolojik Sağlamlık Ölçeği'nin Türkçe uyarlaması: Geçerlik ve güvenirlik çalışması. The Journal of Happiness & Well-Being, 2015; 3(1): 93-102.
- [Background] Jennings-Sanders A. Teaching disaster nursing by utilizing the Jennings Disaster Nursing Management Model. Nurse Educ Pract. 2004 Mar;4(1):69-76. doi: 10.1016/S1471-5953(03)00007-6. PMID 19038139
- [Background] Kalanlar B, Kubilay G. Afetlerde Toplum Sağlığının Korunmasında Önemli Bir Kavram: Afet Hemşireliği. Florence Nightingale Hemşirelik Dergisi, 2015; 23: 57-65
- [Background] Kashiwaba E, Okudera M. Effectiveness of disaster volunteer training as part of basic nursing education. Bulletin of the Faculty of Social Welfare, Iwate Prefectural University, 2014; 16: 1-9.
- [Background] Koca B, Cagan O, Ture A. Validity and reliability study of the Turkish version of the Disaster Response Self-Efficacy Scale in undergraduate nursing students. Acıbadem University Journal of Health Sciences, 2020; 11(3): 515-521. DOI: 10.31067/0.2020.301
- [Background] Inal E, Altintas K. H, Dogan N. The development of a General Disaster Preparedness Belief Scale using the health belief model as a theoretical framework. International Journal of Assessment Tools in Education, 2018; 5: 146-158. doi: 10.21449/ijate.366825
- [Background] Tomizawa Y, Onogi H, Sugawara N, Sugiyama T, Sugawara C, Kawamura M., ... ;Kadoya, K.. Nursing students' learning through volunteer activities after the Great East Japan Earthquake. Bulletin of Tohoku Fukushi University, 2014; 38: 199-220
- [Background] Schmidt CK, Davis JM, Sanders JL, Chapman LA, Cisco MC, Hady AR. Exploring nursing students' level of preparedness for disaster response. Nurs Educ Perspect. 2011 Nov-Dec;32(6):380-3. doi: 10.5480/1536-5026-32.6.380. PMID 22235694
- [Background] Smithers B, Tenhunen ML. Planning and Implementing Disaster Drills for Undergraduate Nursing Students. Nurs Educ Perspect. 2020 Mar/Apr;41(2):130-131. doi: 10.1097/01.NEP.0000000000000430. PMID 30407991
- [Background] Satoh M, Iwamitsu H, Yamada E, Kuribayashi Y, Yamagami-Matsuyama T, Yamada Y. Disaster Nursing Knowledge and Competencies Among Nursing University Students Participated in Relief Activities Following the 2016 Kumamoto Earthquakes. SAGE Open Nurs. 2018 Oct 30;4:2377960818804918. doi: 10.1177/2377960818804918. eCollection 2018 Jan-Dec. PMID 33415208